CLINICAL TRIAL: NCT06576258
Title: The Clinical Impact of Cobas® Eplex Blood Culture Panels for the Diagnosis of Bacteremia and Fungemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EGDE-3742
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-08

CONDITIONS: Bloodstream Infection
Keywords: syndromic diagnostic testing; bloodstream infection; cobas eplex
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention group (eplex implementation) (Experimental): Positive blood culture samples from the intervention group are subjected to eplex multiplex PCR in addition to the SOC culture methods. cobas® eplex system with syndromic panels is a medical device designed for in vitro diagnostic use and is CE-IVD registered. The medical device is used in accordance with the terms of the CE mark.
  Interventions: Diagnostic Test: cobas eplex multiplex PCR

INTERVENTIONS:
Diagnostic Test: cobas eplex multiplex PCR — Positive blood culture samples from the intervention group are subjected to cobas eplex multiplex PCR in addition to the SOC culture methods.

SUMMARY:
A quality improvement study on the diagnostics and clinical management of bloodstream infection episodes. Patients of all ages and genders with positive blood cultures collected for standard patient care are included in the study. In the intervention group of patients, positive blood cultures will be analysed with the cobas® eplex (Roche) blood culture panels in addition to conventional, standard-of-care (SOC) culture methods. The control group will include patients with positive blood cultures analysed using conventional, standard-of-care (SOC) culture methods. The study aims to determine the effect of rapid molecular testing using the cobas® eplex blood culture panels (Roche) in the clinical management of bloodstream infections and more specifically the effect of the eplex result on the time to most effective/targeted antibiotic treatment. The primary objective is to investigate the difference in time to most effective antibiotic treatment between the control and intervention group. The secondary aims are to analyze the concordance of results and compare the user-friendliness, hands-on time and turnaround times of the eplex to the SOC culture methods as well as to compare the difference in the length of stay, antibiotic intensity score at 96h after Gram staining and patient outcome (30-day, all cause mortality and 30-day readmission) in the control and intervention group.

DETAILED DESCRIPTION:
Bloodstream infections (BSIs) impose a considerable burden on patients and healthcare systems due to the need for hospital admission, extended stays, additional diagnostic tests and specific treatments. Receiving inappropriate empirical antibiotic therapy can increase the risk of renal and hepatic toxicity, antibiotic resistance, opportunistic infections and mortality. Therefore, early identification of the causative pathogens and their resistance patterns is of utmost importance.

The gold standard for diagnosis of BSIs is through blood cultures. To detect bacteremia or fungemia, blood from patients is collected and incubated in blood culture bottles. When using conventional culture methods, a positive blood bottle is investigated using direct microscopic investigation, gram-staining, inoculation of selective and non-selective agars, MALDI-TOF identification, rapid antimicrobial susceptibility testing (AST) and standardized AST methods. These methods require several (manual) steps and days of turn-around-time. Following the collection of a blood culture, time to result depends on several factors such as the time needed for transporting the blood bottles and loading in the incubator, the growth rate of bacteria or fungi as well as the time to obtain the identification and AST result.

Rapid diagnostic tests to improve the time to appropriate antimicrobial therapy have been developed. Most tests involve organism identification and genotypic resistance profiles. Rapid molecular diagnostic testing, such as multiplex PCR methods, enable early identification of bacteria or fungi and their antimicrobial resistance genes (results within less than 2 hours after initiation of the test). This helps minimize the time needed to initiate effective antimicrobial therapy. Commercial diagnostic systems to accelerate the identification and detection of antibiotic resistance genes of causative pathogens in BSI have been developed. Examples include Cepheid® GeneXpert, BioFire® FilmArray®TM, and Roche eplex®. The system used in this study, the eplex system, is a random access multiplex PCR platform combining extraction of nucleic acids and rapid RT-PCR. Three Blood Culture Identification (BCID) panels are used to identify the disease-causing organisms: Gram-positive panel, Gram-negative panel and Fungal Pathogen panel. These panels are designed to detect 56 different organisms covering 95% of pathogens commonly associated with BSIs and 10 common antibiotic resistance genes.

The objective of this study is to assess the impact of rapid molecular testing on positive blood cultures with the cobas® eplex system (Roche) on antibiotic therapy and patient outcome.

In this study, we prospectively evaluate the performance of the eplex system for pathogen identification and detection of resistance markers compared to routine SOC for bloodstream infections. The potential impact of the eplex on time to optimization (inititiation, discontinuation, escalation or de-escalation) of antimicrobial therapy and patient outcome will be evaluated.

In summary, Finally, this study will evaluate the potential benefits of implementing CE-IVD registered syndromic diagnostic testing of bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with onset of BSI at the emergency department or general wards
* Patients hospitalized from blood draw (at least 24h)
* For pediatric patient only BSI episodes caused by gram-negative organisms

Exclusion Criteria:

* Patients deceased at the time of the positive blood culture
* Patients in comfort care or with an estimated survival before sepsis of less than one month
* Patients with positive blood culture bottles within the past 14 days
* Patients for which the blood bottles are highly suspected of contaminants (bacterial species belonging to potential skin commensals or known environmental contaminants) and in the absence of any other site of infections.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The time to most effective antimicrobial treatment | From hospital admission until 30 days after discharge of the patient
  The difference in time to most effective/targeted antimicrobial treatment in the intervention group and control group.
  An antimicrobial therapy is defined as optimal when it is the narrowest spectrum agent with acceptable activity against the isolated pathogen based on the culture or eplex results, taking into account the toxicity of the antibiotic and the patient medical conditions.

SECONDARY OUTCOMES:
Performance of the cobas eplex instrument | From positive blood culture until eplex (up to a few hours) and SOC culture results (up to two weeks) are available
  Determine the agreement of the eplex and routine SOC culture results (sensitivity/specificity).
  Determination of user-friendliness and hands-on time of the cobas eplex system. Determination of time-to-result of the eplex compared to routine culture. The time of the eplex identification result is compared to the MALDI-TOF result obtained by the SOC culture method. The time of the eplex AST result is compared to the standardized AST result that is obtained by the SOC culture methods.
The impact of the eplex result on the time to first antibiotic optimization | From hospital admission until the time of first optimization of antimicrobial treatment for the bloodstream infection (up to one week after hospital admission))
  Time to first antibiotic optimization (escalation/de-escalation/change in antibiotic class/discontinuation of therapy) in the control group and the intervention group.
  Definition time to first optimization of antibiotic treatment: the time between the Gram stain result and the first optimization of antibiotic treatment (escalation/de-escalation/change in antibiotic class/discontinuation or initiation of therapy).
  Definition escalation: corresponds to the start of an effective therapy if none had been started or to broadening the bacterial spectrum of the antibiotic therapy.
  Definition de-escalation: defined as narrowing of the antibacterial spectrum of the antibiotic therapy or the stop of at least one antibiotic.
  Definition change in antibiotic class: change in antibiotic class with a similar spectrum of activity.
The impact of the eplex result on the hospital and ICU length-of-stay | From hospital admission until discharge in a single episode of hospitalization, assessed up to one year
  The hospital and ICU length-of-stay of the control group and the intervention group are compared.
  Definition hospital length-of-stay: time between patient's hospital admission and discharge in a single episode of hospitalization.
  Definition ICU length-of-stay: time between the patient's ICU admission and discharge in a single episode of hospitalization.
The impact of the eplex result on 30-day, all cause mortality | From the start of the BSI episode until 30 days after
  The mean 30-day, all cause mortality rate of the control group and the intervention group is compared.
  Definition 30-day, all cause mortality: Mortality from all causes occurring within 30 days of the start of the BSI episode (first positive blood culture).
The impact of the eplex result on antibiotic intensity score at 96 hours after Gram staining | From hospital admission until 96 hours (day 4) after Gram staining
  The antibiotic intensity scores in the control group and the intervention group are compared.
  Definition antibiotic intensity score: The sum of the number of days the patient received of each antibiotic multiplied by the antibiotic spectrum. This value is used to define antibiotic exposure at 96h after Gram staining.
  An antibiotic spectrum index (ASI) matrix was developed by Gerber et al. (2017). To obtain an aggregate ASI for a patient on a single day, the ASI of all antibiotics prescribed are summed.
The impact of the eplex result on 30-day readmission | From hospitalization during the BSI episode until 30 days after discharge
  The 30-day readmission rates of the control group and intervention group are compared.
  Definition 30-day readmission: The 30-day readmission rate is defined as the number of admissions for bloodstream infections for which there was at least one subsequent hospital admission within 30 days after discharge.

OTHER OUTCOMES:
The impact of the eplex result on the health care costs | From hospital admission until discharge in a single episode of hospitalization, assessed up to one year
  Use of health economics models to determine the potential difference in cost based on the length of stay, 30-day all-cause mortality and duration of antimicrobial treatment in the control group and the intervention group.
The impact of the eplex result on patient management | From enrolment until discharge, assessed up to one year
  Determine potential difference in time in patient management between the control group and the study group by monitoring the removal of catheters, additional diagnostic investigations, infection control measures.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Matheeussen, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared. Aggregated patient data will be shared when the findings of the study are made publically available through publication.